CLINICAL TRIAL: NCT01228292
Title: Comparison of Slow Efficiency Daily Dialysis (SLEDD) With Unfractionated Heparin Versus Citrasate in Critically Ill Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Walter Verbrugghe, Critical Care Physician
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/27/179; 2010-021665-68 (EudraCT Number)
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-09

CONDITIONS: Acute Kidney Injury; Hemodialysis
Keywords: Anticoagulation; Intensive Care Medicine; Hemodialysis; Critical Ill Patients
MeSH Terms: conditions — Acute Kidney Injury | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Anticoagulation (Active Comparator): Hemodialysis is performed using standard anticoagulation using unfractionated heparin if no contra-indications for the use of heparin exist. If contra-indications for heparin exist a heparin coated hemofilter (Evodial) will be used. The use of unfractionated heparin or no heparin (with coated hemofilter) is a decision to be taken before every hemodialysis.
  Interventions: Drug: Unfractionated heparin
- Citrasate (Experimental): Hemodialysis is performed with Citrasate
  Interventions: Drug: Citrasate

INTERVENTIONS:
Drug: Unfractionated heparin — dose 5-10 IU/kg/hrs adaptations of infusion rate upon APTT measurements during hemodialysis
  Other Names: Unfractionated Heparin, LEO laboratories Ltd, MA #PL 0043/0041R
  Arms: Standard Anticoagulation
Drug: Citrasate — Citrasate is infused as a dialysate
  Other Names: Citrasate, Advanced Renal Technologies, MA #K000792
  Arms: Citrasate

SUMMARY:
The purpose of this study is to compare the feasibility, safety and efficacy of hemodialysis with unfractionated heparin compared to hemodialysis with Citrasate in Critically Ill Patients.

DETAILED DESCRIPTION:
Objective : To compare the feasibility, safety and efficacy of Sustained Low Efficiency Daily Hemodialysis (SLEDD) using regional anticoagulation with Citrasate® compared to systemic anticoagulation with unfractionated heparin in critically ill patients.

Design : Prospective, randomized, single-center clinical trial Setting : mixed medical-surgical 45 bed ICU in a tertiary university hospital Patients : 250 patients with Acute Kidney Injury (AKI) stage III needing renal replacement therapy Interventions : Patients are randomized to receive SLEDD using standard dialysate and systemic anticoagulation with UF versus SLEDD using Citrasate®-dialysate with no additional UF.

Measurements and main results :

Primary end point :

- The incidence of premature interruptions of the dialysis procedure attributed to hemofilter clotting.

Secondary end points :

* The incidence of bleeding episodes as defined by the WHO-criteria
* The transfusion requirements
* The incidence of technique failure
* The incidence of metabolic derangements (metabolic alkalosis, metabolic acidosis, hypocalcemia, hypercalcemia, hypernatremia, hyponatremia)
* The incidence of citrate intoxication
* The dialysis efficiency expressed as Kt/V and URR

Tertiary end points :

- All cause mortality at day 28 and day 90 after inclusion

ELIGIBILITY:
Inclusion Criteria:

* Need for hemodialysis in the ICU for at least one treatment
* No prior hemodialysis treatment in the ICU except continuous renal replacement therapy

Exclusion Criteria:

* Need for systemic anticoagulation with unfractionated or fractionated heparin, oral anticoagulants or intravenous anti-aggregants for other reasons
* Need for continued thrombolysis therapy within the 6 hours before inclusion
* Need for continued treatment with activated protein C (drotrecogin alfa) within the 12 hours before inclusion
* Need for continued treatment with intravenous anti-aggregants (abciximab, eptifabide) within 12 hours before inclusion
* Liver failure (acute and acute-on-chronic)
* Confirmed or suspected Heparin Induced Thrombocytopenia (HIT)
* Heparin allergies
* Severe uncorrected hypocalcemia (ionized calcium < 0,8 mmol/l)
* Refusal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of premature interruptions of the dialysis procedure attributed to hemofilter clotting. | 6 hours after starting dialysis

SECONDARY OUTCOMES:
The incidence of technique failure defined as the number of patients who develop a contra-indication for the allocated anticoagulation regimen during the study period | during whole wtudy
The incidence of bleeding episodes. A bleeding episode is defined according to the WHO bleeding criteria | during the whole study period
The transfusion requirements defined as the total of units blood products administrated during the ICU stay and per dialysis treatment | during the whole study period
The incidence of metabolic derangements during the study period | during the whole study period
  * Metabolic alkalosis (defined as a pH > 7,5 and a bicarbonate > 24 mmol/l)
  * Metabolic acidosis (defined as a pH < 7,25 and a bicarbonate < 18 mmol/l)
  * Hypocalcemia (defined as an ionized calcium < 0,9 mmol/l)
  * Hypercalcemia (defined as an ionized calcium > 1,2 mol/l)
  * Hypernatremia (defined as a Na+ > 145 mmol/l)
  * Hyponatremia (defined a a Na+ < 130 mmol/l)
  * Citrate toxicity (defined as a total calcium/ionized calcium ratio > 2,5)
Dialysis efficiency expressed as Kt/V and URR | 6 hours after starting dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Karin Jansen-Van doorn, MD, Principal Investigator — Staff member Nephrology Department; Gert Verpooten, PhD, MD, Principal Investigator — Head of Nephrology Department, University Hospital Antwerp, Belgium; Walter Verbrugghe, MD, Principal Investigator — Staff member Critical Care Department, Antwerp University Hospital, Belgium; Philippe Jorens, PhD, MD, Principal Investigator — Head of Critical Care Department, Antwerp University Hospital, Belgium
Locations (1):
- Critical Care Department of the Antwerp University Hospital, Belgium, Edegem, Edegem, Belgium

REFERENCES:
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078